CLINICAL TRIAL: NCT06599112
Title: Clinical and Radiographic Evaluation of Implant Stability in Healed Maxillary Posterior Sites Comparing Osteotome, Osseodensification and Conventional Drilling Implant Placement Techniques: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Implant Stability in Healed Maxillary Posterior Sites Comparing Osteotome, Osseodensification and Conventional Drilling Implant Placement Techniques
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nadine Yehia Mohamed Mohamed Fayed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PERIO631- Perio
Record Dates: First submitted 2024-08-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Implant Stability
Keywords: Dental implant placement; Osseodensification; Osteotomes; Implant stability; Crestal bone loss

STUDY DESIGN:
Intervention Model Description: Three groups. Control Group Intervention group (A) Intervention group (B)
Who Masked: Outcomes Assessor
Masking Description: * Participants and investigator couldn't be blinded.
  * Outcome assessor and biostatistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional drilling for implant placement (Active Comparator): Implant placement in this group will be by conventional drilling according to the manufacturer's instructions (consequent drills according to the kit provided)
  Interventions: Other: Conventional drilling
- Implant placement using Densah Burs (Experimental): Densah Burs provided by Versah will be used as the Osseodensification drilling technique for implant placement in this group. (consequent drilling according to the kit provided)
  Interventions: Other: Densah Burs
- Implant placement using Osteotomes (Experimental): Osteotomes with different serial diameters will be used following the pilot drill to expand and condense the osteotomy site as a technique for implant placement.
  Interventions: Other: Osteotomes

INTERVENTIONS:
Other: Densah Burs — Series of drilling burs inserted in the osteotomy with special design that have a large negative rake angle flute, a cutting chisel edge and a tapered shank, so as they enter deeper into the osteotomy and they have a progressively increasing diameter that controls the expansion process. These burs are used with a standard surgical engine and can densify bone by rotating in the noncutting direction (counterclockwise at 800-1,200 rotations per minute) or drill bone by rotating in the cutting direction (clockwise at 800-1,200 rotations per minute) with an in and out movement together with copious saline irrigation and increasing bone plasticity and ability to expand under rate dependent stress.
  Arms: Implant placement using Densah Burs
Other: Osteotomes — The osteotomes kit are a series of tools that first designed by Summers in 1994. The concept was to maintain the existing bone by compressing trabecular bone laterally and apically with minimal trauma to improve the bone density. The condensed bone in this way will have to put in act a double repairing mechanism, from one side represented by the normal processes of osteointegration and on the other side from the processes of the reparation post fracture like that depends on BMU (bone modelling units) which create new spaces for the new vessels and afterwards filling all the gaps between the bone and the implant.
  Arms: Implant placement using Osteotomes
Other: Conventional drilling — The implant drilling kit provided by the manufacturer will be used for the implant placement, using the pilot drill followed by consequent drills according to the size of the osteotomy needed.
  Arms: Conventional drilling for implant placement

SUMMARY:
This study aims to compare the implant stability values following implant placement via Osteotomes and via Osseodensification using Densah Burs versus implant placement using conventional drilling technique in patients with upper posterior partially edentulous ridges as well as evaluating the crestal bone loss around temporary restorations following the three compared drilling techniques.

DETAILED DESCRIPTION:
* Patients with partially edentulous ridges seeking restoration of their missing teeth, with enough measurements for implant placement will be recruited from the outpatient clinic of the Oral Medicine and Periodontology Department, Faculty of Dentistry-Cairo University to participate in this study and will be randomized to be either undergoing conventional drilling according to the manufacturer's instructions (control group) or either one of the two intervention groups; Intervention group (A) where implant placement will be done using the Osseodensification technique by the Densah burs or Intervention group (B) where the implant placement will be done using the Osteotomes.
* Neobiotech IS III active implants will be used in this study, they have an osseoconductive SLA-coated surface, a tapered design with a crestal macrothread design (0.8 pitch), a self compactable apex as well as deep thread to maximize implant stability. The implant has a platform switching feature and a conical/hex design.
* A temporary PMMA crown after 3 months from implant placement and will be kept for follow up for a year then definitive final restoration will be made.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an age range of 25-70 years
* Patients with systemic health
* Patient with missing teeth in the upper posterior area
* Patients with D3 or D4 type of alveolar bone
* Healed bony sites with sufficient dimension for implant placement

  * Vertical height (≥ 10 mm)
  * Bucco-lingual dimension (≥ 5.5 mm)
  * Mesio-distal width (≥6.5 mm)
* Patients with periodontal health (PD < 4mm, BOP < 10%)
* Inter-arch space of 7.5 to allow implant restoration
* Good oral hygiene
* Cooperative patients who accepted the trial follow up period and sign the informed consent

Exclusion Criteria:

* Pregnant females
* Smokers
* Patients with habits that may compromise the longevity and affect the result of the implant as alcoholism or parafunctional habits
* History of radiotherapy or use of bisphosphonates

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Implant stability. | Will take place at same day,1,2,3,4,6,8 ,12and 16 weeks postoperatively.
  ISQ units. (Implant Stability Quotient)

SECONDARY OUTCOMES:
Crestal bone loss | Will be evaluated to determine the initial crestal bone level at day of the surgery as well at 12 and 48 weeks postoperatively.
  Millimeters in standardized periapical radiograph

OTHER OUTCOMES:
Patient's pain | Same day of surgery as well as 1 week postoperatively.
  Visual Analogue Scale (VAS) on a scale of 0 to 10 where (0) is no pain and (10) is the maximum pain.
Patient satisfaction | Same day f surgery as well as 1 and 2 weeks postoperatively.
  Questionnaire (3 yes or no questions)
Time spent in surgery | Same day of surgery (intraoperatively)
  Minutes using stopwatch.
Patient's pain | Same day of surgery as well as 1 week postoperatively.
  Number of analgesic tablets.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No